CLINICAL TRIAL: NCT04834856
Title: A Phase 2a Open Label, Non-comparative, Single Dose Escalation Study to Evaluate the Dynamics of Viral Clearance, Pharmacokinetics and Tolerability of Ensovibep in Patients With Symptomatic COVID-19 Disease
Brief Title: Viral Clearance, PK and Tolerability of Ensovibep in COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP0420-CP204; 2021-000365-33 (EudraCT Number)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Corona; DARPin
MeSH Terms: conditions — COVID-19 | interventions — ensovibep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ensovibep dose 1 (Experimental)
  Interventions: Drug: ensovibep
- ensovibep dose 2 (Experimental)
  Interventions: Drug: ensovibep

INTERVENTIONS:
Drug: ensovibep — The study will start with a low-dose cohort and after a safety review escalate to the higher dose cohort. One administration at day 1 by infusion.
  Other Names: MP0420

SUMMARY:
This study will investigate how ensovibep is distributed throughout the body, the viral clearance and the tolerability of ensovibep in patients with symptomatic COVID-19 disease

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women, between 18 and 70 years on the day of inclusion.
* Presence of one or more mild or moderate COVID-19 symptoms: Fever, cough, sore throat, malaise, fatigue, headache, muscle pain, gastrointestinal symptoms, or shortness of breath with exertion.
* Positive test for SARS-CoV-2 in upper respiratory swab on the day of dosing (rapid antigen test).

Exclusion Criteria:

* Requiring hospitalization at time of screening, or at time of study drug administration.
* Oxygen saturation (SpO2) ≤ 93 percent (%) on room air at sea level, respiratory rate ≥ 30 per minute, or heart rate ≥125 per minute.
* Any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study.
* Any co-morbidity requiring hospitalization or surgery within <7 days, or that is considered life-threatening within 29 days.
* A patient reported history (prior to the current episode) of a positive SARS-CoV-2 serology test or a history of PCR confirmed SARS-CoV-2 infection.
* Prior or concurrent use of SARS-CoV-2 antiviral medication, including convalescent serum or anti-viral antibodies.
* Concurrent enrollment in any other type of medical research for improving COVID-19 outcomes or that is judged by the investigator not to be scientifically or medically compatible with this study.
* Women that are currently breast feeding, pregnant, or plan to get pregnant during the duration of the trial.
* Severe immunocompromised status (primary immunodeficiency, supraphysiological dose of systemic corticosteroids, transplant patients, known untreated HIV and CD4 T-cells <200/microliter) or use of any immunosuppressants that, in the opinion of the investigator, should preclude participation in this study.
* Subjects at high risk for of COVID-19 related complications or mortality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 viral load | up to day 29
  Changes from baseline to each time point of measurement in SARS-CoV-2 viral load in nasopharyngeal swabs
SARS-CoV-2 viral cultures | up to day 29
  Changes from baseline to each time point of measurement in SARS-CoV-2 viral cultures cultivated from nasopharyngeal swabs
SARS-CoV-2 PCR days to negativity | up to day 29
  Duration in days to SARS-CoV-2 PCR negativity
Observed maximum concentration (Cmax) | up to day 91
  The maximum observed concentration (Cmax) is estimated based on the serum concentrations.
Terminal Elimination Half-Life (T½) | up to day 91
Time to Cmax (Tmax) | up to day 91
The area under the concentration-time curve from time zero extrapolated to infinity time (AUCinf) | up to day 91
The area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | up to day 91
Apparent total body clearance of the drug from plasma (CL) | up to day 91
Apparent volume of distribution at steady state (Vss) | up to day 91

SECONDARY OUTCOMES:
14 Common Covid-19 Related Symptoms score | up to day 29
  Changes in the assessment of 14 Common Covid-19 Related Symptoms score
Treatment-emergent (serious) adverse events ((S)AEs) and AEs of Special Interest (AESIs) including Infusion-related reactions (IRRs) | up to day 91
  Treatment-emergent (S)AEs and AESIs, including infusion-related reactions (IRRs) will be assessed throughout the study
Concomitant medication | up to day 91
  Intake of concomitant medication will be assessed throughout the study
Vital Signs: Heart Rate (bpm) | up to day 91
Vital Signs: Blood Pressure Systolic and Diastolic (mmHg) | up to day 91
Vital Signs: Respiratory Rate (breaths per minute) | up to day 91
Vital Signs: Body Temperature (°C) | up to day 91
Vital Signs: Oxygen Saturation (SpO2) | up to day 91
Clinical laboratory tests (hematology and blood chemistry) | up to day 91
Physical examinations (symptom directed) | up to day 91
Local tolerability at injection site | up to 90 min post dose
  Local tolerability at injection site will be assessed via Visual Infusion Phlebitis score

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands